CLINICAL TRIAL: NCT04235517
Title: Behaviour of the Growth Plate in Patients Operated With Either Permanent or Temporary Hemi-epiphysiodesis or Epiphysiodesis Through by the Use of Radiostereometric Analysis (RSA)
Brief Title: RSA Study on the Behaviour of the Growth Plate During and After Temporary Hemi-epiphysiodesis and Epiphysiodesis
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anne Berg Breen, Principal Investigator, Oslo University Hospital
Other Study IDs: 18/02287
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Anisomelia; Deformity of Limb
Keywords: LLD, guided growth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Axial deviations in children: Children with axial deviations in the lower extremity treated with guided growth
  Interventions: Other: Temporary hemi-epiphysiodesis or epiphysiodesis
- Limb length discrepancy in children: Children with limb length discrepancy treated with temporary epiphysiodesis
  Interventions: Other: Temporary hemi-epiphysiodesis or epiphysiodesis

INTERVENTIONS:
Other: Temporary hemi-epiphysiodesis or epiphysiodesis — Tension band plate (eight-plate, pedi plate), staple or locking plate

SUMMARY:
By using radiostereometric analysis (RSA) we will be able to study growth during and after temporary epiphysiodesis and with great accuracy be able to detect asymmetric growth following this procedure.

By using the same method we also want to analyse patients with axial deviations operated with guided growth (tension band plating) to study the growth during and after the procedure and be able to set the correct timing for removal of the implant.

DETAILED DESCRIPTION:
The RSA method consists of implantation of small tantalum beads on either side of the physis during surgery on the the physis. Later analysis of the RSA Pictures with the RSA-method will give us an microscopically accurate measure of the growth in three planes.

ELIGIBILITY:
Inclusion Criteria:

* Children with idiopathic axial deviations in the lower extremities
* Children with limb length discrepancys where timing of epiphysiodesis is difficult because of a big discrepancy in skeletal age and chronological age

Exclusion Criteria:

* Children with axial deviations and pathological physis

Ages: 3 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Children with growth remaining and limb length discrepancy or axial deviations in the lower extremity
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Behaviour of the growth plate during and after temporary hemi-epiphysiodesis and epiphysiodesis | 4 years
  Radiostereometric analysis of growth

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Horn, MD,PHD, Study Chair — Oslo Unversity Hospital
Locations (1):
- The Ortopedic dep at Oslo Unversity Hospital, Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No